CLINICAL TRIAL: NCT05369325
Title: Accuracy of Non-invasive Hemoglobin Monitoring in Patients Undergoing Outpatient Total Joint Arthroplasty
Brief Title: Non-invasive Hemoglobin Monitoring in Outpatient Total Joint Arthroplasty
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Matthew P. Abdel, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 22-000012
Record Dates: First submitted 2022-05-03; First posted 2022-05-11 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Total Joint Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research is being done to better understand the accuracy of noninvasive hemoglobin tests on patients that recently underwent total joint arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients age ≥ 18.
* Undergoing either primary total knee or total hip arthroplasty for a primary underlying diagnosis of osteoarthritis.

Exclusion Criteria:

- Individuals < 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing total joint arthroplasty at Mayo Clinic
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Concordance between non-invasive Hgb and serum Hgb | 1 hour
  How closely the non-invasive and serum Hgbs correlate with one another statistically
Patient satisfaction with non-invasive Hgb | 1 day
  Patients will get a survey to fill out following the Hgb measurements that assesses their satisfaction with the non-invasive method
Nurse satisfaction with non-invasive Hgb | 1 day
  Nurses will get a survey to fill out following the Hgb measurements that assesses their satisfaction with the non-invasive method
Cost comparison between non-invasive and serum Hgb | 1 year
  We will analyze cost differences between the non-invasive Hgb devices and the serum lab tests

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Abdel, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials